CLINICAL TRIAL: NCT02722733
Title: Safety and Efficacy of Stem Cell Mobilization Using G-CSF (Filgrastim) Alone Compared to Intermediate-dose Cytosine Arabinoside Plus G-CSF in Hodgkin's Lymphoma and Non-Hodgkin's Lymphoma Patients.
Brief Title: Randomized Trial of G-CSF Alone Versus Intermediate-dose Ara-C Plus G-CSF Mobilization in Hodgkin's Lymphoma or Non-Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Responsible Party: Principal Investigator, Sebastian Giebel, Prof., MD, Maria Sklodowska-Curie National Research Institute of Oncology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HL/NHLMobil-COI-01
Record Dates: First submitted 2016-03-11; First posted 2016-03-30 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Hodgkin's Lymphoma; Non-Hodgkin's Lymphoma
Keywords: Hodgkin's lymphoma; Non-Hodgkin's lymphoma; mobilization; G-CSF; filgrastim; cytosine arabinoside; autologous stem cell transplantation
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin | interventions — Granulocyte Colony-Stimulating Factor; Filgrastim; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- G-CSF (filgrastim) (Active Comparator): 1.G-CSF at 10 μg/kg per day (divided into two doses every 12 hours) subcutaneously for up to 7 days.
  Interventions: Drug: G-CSF (filgrastim)
- Cytosine arabinoside + G-CSF (filgrastim) (Active Comparator): 1. Cytosine arabinoside will be administered as a 2-hour i.v. infusion at a dose of 0.4 g/m2 twice daily on days 1 and 2 (total dose 1.6 g/m2).
  2. G-CSF 5-10 μg/kg per day (divided into two doses every 12 hours) will be started on day 5 subcutaneously and continued until last leukapheresis.
  Interventions: Drug: Cytosine arabinoside with G-CSF (filgrastim)

INTERVENTIONS:
Drug: G-CSF (filgrastim)
  Arms: G-CSF (filgrastim)
Drug: Cytosine arabinoside with G-CSF (filgrastim)
  Arms: Cytosine arabinoside + G-CSF (filgrastim)

SUMMARY:
The purpose of the study is to compare safety and efficacy of stem cell mobilization using G-CSF (filgrastim) alone vs. intermediate-dose cytosine arabinoside plus G-CSF in Hodgkin's lymphoma and non-Hodgkin's lymphoma patients.

DETAILED DESCRIPTION:
Autologous hematopoietic stem cell transplantation (autoHSCT) is a standard treatment of eligible patients suffering from Hodgkin's Lymphoma or non-Hodgkin's Lymphoma (HL, NHL). AutoHSCT allows to further improve results of the therapy. Nowadays, 99% of the procedures are performed using peripheral blood as a source of stem cells. Hence, the crucial point is to harvest adequate number of stem cells allowing hematopoietic recovery. The number of 2 × 10^6 CD34+ cells/kg is considered the minimal level in autoHSCT. There are two main mobilization strategies being used: based on G-CSF alone or in combination with chemotherapy (cyclophosphamide (CY) at dose range 1.6 g/m2 is mainly used in HL and NHL setting). However, a proportion of patients (5-40%) fail to collect the minimum number of cells required. Novel agents, like plerixafor, CXCR4 inhibitor, may enable effective CD34+ cell harvest in "poor mobilizers". Nevertheless, the optimal first-line and cost-effective protocol for mobilization of hematopoietic stem cells has not been determined so far.

Randomized trials compare chemomobilization with the use of CY + G-CSF to G-CSF alone, which had been conducted so far, did not demonstrate clear advantage of addition of CY to the growth factor. Intermediate-dose cytosine arabinoside (AraC), 1.6 g/m2 plus filgrastim, has been shown to produce very high efficacy as a first or second-line mobilization regimen in patients with lymphoid malignancies. In a retrospective comparison, this strategy was significantly more effective than CY + G-CSF. This suggest that the type of chemotherapy agent added to G-CSF may play role in mobilization efficacy and that the combination of AraC and G-CSF may be more effective than G-CSF used alone. The goal of current study is to verify this hypothesis in randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. Hodgkin's lymphoma and non-Hodgkin's lymphoma patients considered eligible for autologous stem cell transplantation procedure.
2. Must not have achieved complete remission after first line of therapy or must have relapsed lymphoma.
3. Must have received at least two lines of therapy including four or more cycles.
4. Must have achieved a partial (PR) or complete remission (CR) .
5. Must be 18-65 years of age.
6. Must have World Health Organization performance status 0-1.
7. Time from administration or discontinuation of any chemotherapy agent must be at least four weeks.
8. Hemoglobin level > 8 g/dl, Absolute neutrophil count (ANC) > 1.5 x 10^9/L, Platelet count >100 x 10^9/L.
9. Serum creatinine < 1.5 x upper limit of normal (ULN), serum bilirubin < 1.5 ULN, serum aspartate transaminase (AST/SGOT) < 2.5 x ULN, serum alanine transaminase (ALT/SGPT) < 2.5 x ULN.
10. Negative human immunodeficiency virus (HIV) infection test.
11. Negative pregnancy test.
12. Must understand and voluntarily sign informed consent form.

Exclusion Criteria:

1. Failure of prior, first-line mobilization regimen.
2. Infiltration of central nervous system.
3. Bone marrow plasma cell infiltration of above 20%.
4. Administration of nitrosourea derivatives (Carmustine, Lomustine) within 4 weeks before starting study treatment.
5. Administration of growth-factor other than G-CSF Administration of G-CSF within 14 days before starting study treatment.
6. Ongoing or active infection.
7. Coexisting neoplasm, other than Hodgkin's or non-Hodgkin's lymphoma.
8. Administration of radioimmunotherapy in past.
9. Pregnant or lactating females.
10. Patients treated with use of autologous or allogenic stem cell transplantation in the past.
11. Positive human immunodeficiency virus (HIV) infection test.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
• The proportion of patients with stem cell yield at least 2 × 10^6 CD34+ cells/kg in each treatment arm. | After up to three leukaphereses (7-20 days after starting mobilization regimen).

SECONDARY OUTCOMES:
Peak level of CD34+ cells in peripheral blood (cells/μl). | 7-20 days after starting mobilization regimen.
Total number of harvested CD34+cells/kg. | After up to three leukaphereses (7-20 days after starting mobilization regimen).
Number of leukaphereses needed to harvest target amount of stem cells. | 7-20 days after starting mobilization regimen.
The proportion of hematologic and non-hematologic complications. | 1 month after transplantation.
Duration of neutropenia < 0.5 x10^9/L. | 1 month after transplantation.
Number of blood transfusions needed. | 1 month after transplantation.
Duration of hospital stay. | 1 month after transplantation.
Time of neutrophil and platelet engraftment after autologous stem cel transplantation. | 1 month after transplantation.
Duration of thrombocytopenia <50 x 10 ^9/L. | 1 month after transplantation.
Number of days of antibiotics therapy. | 1 month after transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Gliwice Branch, Gliwice, Poland

REFERENCES:
- [Background] Narayanasami U, Kanteti R, Morelli J, Klekar A, Al-Olama A, Keating C, O'Connor C, Berkman E, Erban JK, Sprague KA, Miller KB, Schenkein DP. Randomized trial of filgrastim versus chemotherapy and filgrastim mobilization of hematopoietic progenitor cells for rescue in autologous transplantation. Blood. 2001 Oct 1;98(7):2059-64. doi: 10.1182/blood.v98.7.2059. PMID 11567990
- [Background] Karanth M, Chakrabarti S, Lovell RA, Harvey C, Holder K, McConkey CC, McDonald D, Fegan CD, Milligan DW. A randomised study comparing peripheral blood progenitor mobilisation using intermediate-dose cyclophosphamide plus lenograstim with lenograstim alone. Bone Marrow Transplant. 2004 Sep;34(5):399-403. doi: 10.1038/sj.bmt.1704598. PMID 15273706
- [Background] Sheppard D, Bredeson C, Allan D, Tay J. Systematic review of randomized controlled trials of hematopoietic stem cell mobilization strategies for autologous transplantation for hematologic malignancies. Biol Blood Marrow Transplant. 2012 Aug;18(8):1191-203. doi: 10.1016/j.bbmt.2012.01.008. Epub 2012 Jan 16. PMID 22261379
- [Background] Kruzel T, Sadus-Wojciechowska M, Najda J, Czerw T, Glowala-Kosinska M, Holowiecki J, Giebel S. Very high efficacy of intermediate-dose cytarabine in combination with G-CSF as a second-line mobilization of hematopoietic stem cells. Int J Hematol. 2012 Aug;96(2):287-9. doi: 10.1007/s12185-012-1135-5. Epub 2012 Jul 14. No abstract available. PMID 22797877
- [Background] Giebel S, Kruzel T, Czerw T, Sadus-Wojciechowska M, Najda J, Chmielowska E, Grosicki S, Jurczyszyn A, Pasiarski M, Nowara E, Glowala-Kosinka M, Chwieduk A, Mitrus I, Smagur A, Holowiecki J. Intermediate-dose Ara-C plus G-CSF for stem cell mobilization in patients with lymphoid malignancies, including predicted poor mobilizers. Bone Marrow Transplant. 2013 Jul;48(7):915-21. doi: 10.1038/bmt.2012.269. Epub 2013 Jan 7. PMID 23292239